CLINICAL TRIAL: NCT03424486
Title: Prevalence and Impact of Depression and Anxiety in Cystic Fibrosis
Acronym: ADMPE-2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Other Study IDs: NI17007JJ
Record Dates: First submitted 2017-11-17; First posted 2018-02-07 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Anxiety; Depression; Adolescence
MeSH Terms: conditions — Cystic Fibrosis; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents (14 to 17 years old): Patients with CF
  Interventions: Other: Questionnaires
- Parents: Parents of adolescents (14 to 17 years old with CF (father, mother and other)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Evaluation of the prevalence of anxiety, depression and quality of life

SUMMARY:
The Impact of cystic fibrosis (CF) on psychological and emotional functioning has been the focus of several studies over the past 20 years. The results from a current meta-analysis indicated that depressed patients were three times more likely to be noncompliant with treatment recommendations than nondepressed patients with chronic illness.

To date, most studies of the prevalence of psychiatric symptoms have been limited by small sample size; reliance on samples of convenience that are potentially biased in term of rates of symptomatology, and measures that contain legitimate symptoms that are part of the respondent's chronic disease. Estimating the prevalence of depression and anxiety has become important as new evidence indicates that these symptoms may have a significant impact on health outcomes, including adherence to medical treatments, utilization of health care services, and rates of morbidity and mortality. More depressive the symptoms are associated with poorer lung function, and that in the absence of depression, poor lung function is minimally associated with lower patient ratings of quality of life.

The purpose of the current study is to estimate the regional, and if possible the national prevalence of depressive and anxious symptoms in children and adults with CF and parents caregivers. Patients with CF ages 14 to 17, and parents of children ages 14 to 17, will complete and depression/anxiety screening measure at a routine clinic visit. These will then be linked with demographic and medical variables reported to the CF registry and analyzed cross sectionally. Adults with CF ages 18 and older will also complete the depression / anxiety screening measure at a routine clinic visit. Efforts will be made to recruit a representative sample of patients from each clinic.

DETAILED DESCRIPTION:
Numerous studies have demonstrated that patients with chronic illnesses are at increased risk for depression and anxiety. In large, well-controlled epidemiological studies, rates of depression in medical populations have ranged from 17% to 50% compared to 5% to 17.5% in healthy populations. Reporting on a community-based sample, Wells and colleagues concluded that individuals with a chronic medical condition have a 41% increase in the risk of having a psychiatric disorder as well.

In patients with chronic illnesses, depression and anxiety have been shown to have direct and indirect consequences for health outcomes, and this has been addressed in a recent ATS/ERS consensus statement on pulmonary rehabilitation. Depressed patients are less compliant with medical regimens, less likely to follow dietary regimes, more likely to cancel or miss clinic appointments, report worse functioning on several quality of life domains, have increased health care utilization and higher health care costs, and are also more likely to engage in risky behaviors, such as smoking, drinking and drug use.

To date, studies of the impact of depression and anxiety in patients with CF have been limited by small samples sizes, samples of convenience that may provide biased estimates of symptom rates, and have used measures that confound symptoms of depression with those of a chronic illness. Given the importance of identifying and treating these symptoms, and their implications for long-term health outcomes, the current study proposes to conduct the first national prevalence study of depression and anxiety in CF patients and parent caregivers. Furthermore, we plan to examine the impact of these psychological symptoms on health outcomes, such as pulmonary exacerbations and nutritional status.

1. Anxiety and Depression are common in Cystic Fibrosis, but their exact prevalence is unknown.

   Specific Aim 1: To estimate the prevalence of depression and anxiety in patients with CF ages 14 to 17 and parent caregivers of those adolescents

   Of the few studies of school-age children and adolescents with CF, one reported a rate of depression ranging from 11% to 14.5% in contrast to a rate of 2-6% in the general pediatric population. Published rates of anxiety have ranged from 5% to 9% which may approximate that of the general childhood population. Furthermore, the rate of depression in parent caregivers is also high compared to parents of healthy children. In a multi-site adherence intervention trial of 88 parents of young children with CF, ages 1 to 11, 29% of parents scored in the clinical range on a depression screening tool. This is similar to a study of role strain in parents of young children with CF, in which 36.4% of the mothers' depressive symptoms fell within the clinical range. Furthermore, even higher rates of depression were reported in a study of parents soon after the diagnosis, with 64% of mothers and 43% of fathers scoring in the clinical range.

   Previous estimates of the prevalence of depression and anxiety in patients with CF have been hampered by serious methodological limitations, such as small sample size, convenience sampling that is potentially biased, and the use of diagnostic screening instruments that attribute somatic symptoms to a depressive disorder which may be due to having a chronic illness like CF (e.g., fatigue). Furthermore, studies of depression and anxiety in pediatric CF populations have not considered developmental and gender differences in depression that emerge in the general population during adolescence.
2. Identifying patients and parents at risk for depression and anxiety disorders is important, but risk factors in the CF population are not known.

   Specific Aim 2: To identify risk factors associated with symptoms of depression and anxiety.

   This study was cross-sectional, making it impossible for the authors to distinguish whether psychological symptoms preceded or followed patients' employment status, or how either of these might have been related to changes in health outcomes.
3. Anxiety and depression probably lead to worse clinical outcomes in CF, but this has not been evaluated.

Specific Aim 3: To evaluate how depression and anxiety influence health outcomes (particularly number of exacerbations and hospitalizations, FEV1 and nutritional measures) over the ensuing year.

There is wide variability in the progression of disease in patients with CF, as reflected in the distribution of age at diagnosis, age-related pulmonary function, and age at death (Cystic Fibrosis Foundation Patient Registry, 2004). This variability is partially explained by CFTR mutation and gene modifiers, but environmental and sociodemographic factors, and variations in the use of various healthcare interventions are of equal or greater importance in explaining this variability in health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CF
* 14 to 17 year old
* Parents of a included patient

Exclusion Criteria:

- Patient who have received an organ transplant shall be excluded.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Patients with CF aged 14 to 17. Patients awaiting organ transplantation will be included in the study, but those who have received an organ transplant shall be excluded. No other exclusionary criteria will be used.
  2. Parents of the patients included.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression in patients with CF ages 14 to 17 and their parent caregivers | at inclusion (1 day)
  The depression is assessed with the HADS scale (Hospital Anxiety and Depression Scale) at the inclusion (Day 1) : the depression HADS score [0-21]

SECONDARY OUTCOMES:
Identification of the risk factors associated with symptoms of depression | at the inclusion (1 day)
  Symptoms of depression are assessed with the Center for Epidemiological Studies of Depression Scale (CES-D) : CES-D score [0-60]
Identification of the risk factors associated with symptoms of anxiety | at the inclusion (1 day)
  The anxiety is assessed with the HADS scale : the anxiety HADS score [0-21]
Measure of the Quality of life of adolescents with CF (14-17) | at the inclusion (1 day)
  The quality of life of adolescents is assessed with the Cystic Fibrosis Questionnaire (CFQ14+) : CFQ score
Change in FEV1 over the ensuing year | 12 months
  FEV1 (in % predicted)
Change in BMI over the ensuing year | 12 months
  Weight (Kg) and height (m) will be combined to report BMI in kg/m2
Number of exacerbations over the ensuing year | 12 months
  Number of exacerbations over the 12 last months to identify the risk factors associated with symptoms of depression and anxiety, and to evaluate the influence of depression and anxiety on CF health outcomes
Number of hospitalizations over the ensuing year | 12 months
  Number of hospitalizations over the 12 last months to identify the risk factors associated with symptoms of depression and anxiety, and to evaluate the influence of depression and anxiety on CF health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: MAYA KIRSZENBAUM, MsD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (8):
- France (8):
  - CRCM - Service de Pneumologie Pédiatrique - CHU Amiens - Site Sud, Amiens
  - CRCM Enfants - Service de Pneumologie - Hôpital Jean Minjoz, Besançon
  - CRCM Pédiatrique - Hôpital des Enfants, Bordeaux
  - CRCM - Service de Pédiatrie - Pôle FEH - CHU Caen), Caen
  - CRCM / Service de Médecine Infantile - Hôpital d'Enfants - CHRU Nancy, Nancy
  - Department of Pneumology - CRCM- Necker - Enfants malades Hospital (AP-HP) -, Paris
  - CRCM - Service de Pédiatrie A - American Memorial Hospital, Reims
  - CRCM / Service de Pédiatrie _ Hôpital de Clocheville - CHRU de Tours, Tours